CLINICAL TRIAL: NCT06049745
Title: Use of Misoprostol in Hysteroscopic Myomectomy, a Randomized Peospective Trial
Brief Title: Use of Misoprostol in Hysteroscopic Myomectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Collaborators: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Oshri Barell, Head of Gynecology Division, Department of Obstetrics and Gynecology. Assuta Ashdod University Hospital, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0083-23-AAA
Record Dates: First submitted 2023-08-29; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hysteroscopic Myomectomy
Keywords: hysteroscopic myomectomy; misoprostol

STUDY DESIGN:
Intervention Model Description: patients undergoing hysteroscopic myomectomy will be divided into two groups, the study group will receive misoprostol before the procedure. the control group will not receive treatment with misoprostol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hysteroscopic myomectomy without misoprostol (No Intervention): Patients undergoing hysteroscopic myomectomy that will be randomized to no intervention before the procedure.
- Misoprostol group (Experimental): Patients undergoing hysteroscopic myomectomy will be randomized to 400 mcg of misoprostol sublingual before the procedure.
  Interventions: Drug: Misoprostol 400 Microgram Oral Tablet

INTERVENTIONS:
Drug: Misoprostol 400 Microgram Oral Tablet — S.L misoprostol 400 mcg
  Arms: Misoprostol group

SUMMARY:
Hysteroscopic myomectomy is typically suitable for myomas measuring under 4 cm in size. The utilization of misoprostol before the procedure can facilitate uterine access, decrease fluid absorption, and reduce blood loss, consequently leading to a decrease in the overall procedure time. In this randomized trial, the investigators aim to investigate the impact of misoprostol administration and its effects on each of the mentioned parameters.

DETAILED DESCRIPTION:
Hysteroscopic myomectomy is a minimally invasive surgical procedure designed to remove uterine fibroids that are located within the uterine cavity. Traditionally, hysteroscopic myomectomy for large fibroids has been performed as a two-step procedure, with fibroid removal divided into separate stages. However, advancements in surgical techniques and equipment have allowed for the development of hysteroscopic myomectomy as a one-step procedure, in which all fibroids are removed in a single surgical session.

As a one-step procedure, hysteroscopic myomectomy offers several potential benefits. It eliminates the need for multiple surgeries and reduces the overall treatment timeline for patients. The size limit for hysteroscopic myomectomy varies among surgeons and institutions. In general, submucosal fibroids up to 4 centimeters in diameter are considered suitable for hysteroscopic resection.

Fluid overload is an important consideration in hysteroscopic myomectomy, especially when it is performed as a one-step procedure, making it a time-limited procedure. During hysteroscopic myomectomy, a distension media is used to expand the uterine cavity, providing better visualization and creating a working space for the surgeon. However, there is a risk of fluid overload if excessive fluid is absorbed into the bloodstream, potentially leading to complications such as electrolyte imbalances, fluid imbalance, hyponatremia, or cardiovascular issues. To mitigate this risk, certain precautions are taken during the procedure.

When the uterus contracts, the fibroid may undergo several changes. These changes can affect the position, size, and accessibility of the fibroid, potentially influencing the surgical approach and outcome. Fibroid extrusion occurs when the fibroid becomes detached from its attachment site and is pushed out of the uterus by the uterine contractions.

A case study published by Murakami et al. discussed the contributing effect of intraoperative injection of prostaglandin F2 alpha in a patient undergoing hysteroscopic myomectomy, resulting in a successful one-step hysteroresectoscopy of a sessile submucous leiomyoma . Additionally, Indman described the effect of intracervical injection of carboprost prior to hysteroscopic resection of submucous myomas that could not be completely resected in a series of 10 case studies .

To the investigators knowledge, the use of misoprostol in hysteroscopic resection has been primarily limited to its role as a cervical dilation primer prior to the procedure. The use of misoprostol in hysteroscopy may reduce the need for mechanical cervical dilatation , however, many centers do not use misoprostol routinely in every hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* women between the ags of 20 years- 55 years, inclusive
* undergoing hysteroscopic myomectomy
* submucosal fibroid less than 40 mm (type 0, 1 and 2)
* up to 2 submucosal fibroids
* patients are able to provide written informed consent

Exclusion Criteria:

* post menopausal women
* inability to perform operative hysteroscopy under anesthesia in the past due to cervical stenosis
* previous PID or documented tubal occlusion
* positive BHCG test
* inability to consent due to cognitive or language barrier
* allergy to misoprostole
* severe COPD, asthma or cardiac disease

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
length of the procedure | from the first insertion of the hysteroscope to the end of the procedure, minutes
  overall procedure time

SECONDARY OUTCOMES:
fluid absorption | from the start of the procedure to the end of the procedure
  fluid deficit as measured within the procedure
success in one procedure | from the start of the procedure to the end of the procedure
  complete removal of the fibroid in a one step procedure
surgical complications | 1 month folowing the procedure
  surgical complications according to the Dindo-Clavien scale
patient satisfaction | within 30 days of the procedure
  satisfaction from the procedure on a scale of 1-10
blood loss | from the start of the procedure until the patient has left the operating room
  estimated blood loss as measured by the surgeon during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moawad NS, Palin H. Hysteroscopic Myomectomy. Obstet Gynecol Clin North Am. 2022 Jun;49(2):329-353. doi: 10.1016/j.ogc.2022.02.012. PMID 35636812
- [Background] Loddo A, Djokovic D, Drizi A, De Vree BP, Sedrati A, van Herendael BJ. Hysteroscopic myomectomy: The guidelines of the International Society for Gynecologic Endoscopy (ISGE). Eur J Obstet Gynecol Reprod Biol. 2022 Jan;268:121-128. doi: 10.1016/j.ejogrb.2021.11.434. Epub 2021 Dec 1. PMID 34902749
- [Background] Zayed M, Fouda UM, Zayed SM, Elsetohy KA, Hashem AT. Hysteroscopic Myomectomy of Large Submucous Myomas in a 1-Step Procedure Using Multiple Slicing Sessions Technique. J Minim Invasive Gynecol. 2015 Nov-Dec;22(7):1196-202. doi: 10.1016/j.jmig.2015.06.008. Epub 2015 Jun 18. PMID 26093183
- [Background] Indraccolo U, Bini V, Favilli A. Likelihood of Accomplishing an In-Patient Hysteroscopic Myomectomy in a One-Step Procedure: A Systematic Review and Meta-Analysis. Biomed Res Int. 2020 Jan 8;2020:4208497. doi: 10.1155/2020/4208497. eCollection 2020. PMID 32090092
- [Background] Umranikar S, Clark TJ, Saridogan E, Miligkos D, Arambage K, Torbe E, Campo R, Di Spiezio Sardo A, Tanos V, Grimbizis G; British Society for Gynaecological Endoscopy /European Society for Gynaecological Endoscopy Guideline Development Group for Management of Fluid Distension Media in Operative Hysteroscopy. BSGE/ESGE guideline on management of fluid distension media in operative hysteroscopy. Gynecol Surg. 2016;13(4):289-303. doi: 10.1007/s10397-016-0983-z. Epub 2016 Oct 6. No abstract available. PMID 28003797
- [Background] Murakami T, Shimizu T, Katahira A, Terada Y, Yokomizo R, Sawada R. Intraoperative injection of prostaglandin F2alpha in a patient undergoing hysteroscopic myomectomy. Fertil Steril. 2003 Jun;79(6):1439-41. doi: 10.1016/s0015-0282(03)00386-8. PMID 12798895
- [Background] Indman PD. Use of carboprost to facilitate hysteroscopic resection of submucous myomas. J Am Assoc Gynecol Laparosc. 2004 Feb;11(1):68-72. doi: 10.1016/s1074-3804(05)60014-x. PMID 15104835
- [Background] Al-Fozan H, Firwana B, Al Kadri H, Hassan S, Tulandi T. Preoperative ripening of the cervix before operative hysteroscopy. Cochrane Database Syst Rev. 2015 Apr 23;2015(4):CD005998. doi: 10.1002/14651858.CD005998.pub2. PMID 25906113
- [Background] Lasmar RB, Lasmar BP, Celeste RK, da Rosa DB, Depes Dde B, Lopes RG. A new system to classify submucous myomas: a Brazilian multicenter study. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):575-80. doi: 10.1016/j.jmig.2012.03.026. Epub 2012 Jul 20. PMID 22819007